CLINICAL TRIAL: NCT01313897
Title: UARK 2010-35, A Phase II Study of Expanded Natural Killer Cell Therapy for Multiple Myeloma
Brief Title: UARK 2010-35, A Study of Expanded Natural Killer Cell Therapy for Multiple Myeloma
Acronym: NK2010-35
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 114344; IND 14560 (Other: Food and Drug Administration)
Record Dates: First submitted 2010-12-01; First posted 2011-03-14 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Velcade for Anti-MM therapy (Experimental): Day(s) -9,-6,-2 3 doses of Bortezomib at 1.0 mg/m2, i.v.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — bortezomib to be given days -9, -6, and -2 at 1.0mg/m2, i.v.
  Other Names: Velcade

SUMMARY:
The purpose of this study is to determine the therapeutic efficacy of the exp-NK cell therapy in research participants with relapsed high risk MM [defined as gene expression profile (GEP) 70 gene score ≥0.66 and/or metaphase chromosomal abnormalities and/or high LDH ≥ 360U/L] by establishing the (near) complete response rate. Response rate will be compared to case matched historical controls (patients who relapsed on Total Therapy 2 or 3 with high-risk MM defined as above). Disease-free survival and overall survival will be captured but are not primary or secondary endpoints.

DETAILED DESCRIPTION:
The use of auto-exp-NK cells in this protocol makes therapy available to all refractory high risk MM patients, 2/3 of whom would otherwise not have a suitable haploidentical donor. We have shown that NK cells can be expanded both from newly diagnosed high risk MM patients and from refractory, previously heavily treated patients, the very individuals in need of novel therapies such as exp-NK cell infusions. Furthermore, we observed that exp-NK cells have the ability to kill auto-MM cells in vitro compared to no killing with resting auto-NK cells. This may be due to the elevated activation state of exp-NK cells, which allows them to overcome otherwise dominant inhibitory signaling. The incorporation of the proteasome inhibitor bortezomib, which down regulates the principal NK cell inhibitory ligands on MM cells should further increase the efficacy of auto-exp-NK cells. Because there is no risk for GvHD, CD3+ T cell depletion will not be necessary for auto-exp-NK cell products.

ELIGIBILITY:
Inclusion Criteria:

* Patient (Recipient of NK Cells) Inclusion Criteria
* Relapsed patients must have high risk disease as defined by GEP risk score of ≥ 0.66 or metaphase cytogenetic abnormalities or LDH ≥ 360 U/L (Rule out hemolysis, infection and contact PI for clarification if any doubt) Patients must have had at least 1 line of prior chemotherapy and/or have relapsed after auto- PBSCT.
* For subjects who have had a prior transplant, ≥2 months must have relapsed after the last transplant prior to enrollment.
* Zubrod ≤ 2, unless solely due to symptoms of MM-related (bone) disease.
* Patients must have a platelet count of ≥ 50,000/µL within 35 days of registration, unless lower levels are explained by extensive bone marrow plasmacytosis or extensive prior therapy.
* Patients must be at least 18 years of age and not older than 75 years of age at the time of registration.
* Participants must have preserved renal function as defined by a serum creatinine level of ≤ 3 mg/dL within 35 days of registration.
* Participants must have an ejection fraction by ECHO or MUGA scan ≥ 40% within 90 days prior to registration.
* Patients must have adequate pulmonary function studies > 50% of predicted on mechanical aspects (FEV1, FVC, etc) and diffusion capacity (DLCO) > 50% of predicted within 90 days prior to registration. If the patient is unable to complete pulmonary function tests due to MM related pain or condition, exception may be granted if the principal investigator documents that the patient is a candidate for high dose therapy.
* Patients must have signed an IRB-approved informed consent and HIPAA authorization form.
* Either a haploidentical family donor fit to undergo leukapheresis is available or the recipient is fit to undergo leukapheresis for exp-NK cell generation (see donor selection).
* Patient (Recipient of NK Cells) Exclusion criteria
* History of poorly controlled hypertension, diabetes mellitus, or any other serious medical illness or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol or could be considered to be an exclusion criterion deemed by the PI.
* Patients must not have prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has not received treatment for one year prior to enrollment. Other cancers will only be acceptable if the patient's life expectancy exceeds three years as determined by the PI.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of registration. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Donor Inclusion Criteria
* The source of the NK cells will be either A) a family member who is HLA haploidentical to the recipient, or B) if a suitable haploidentical donor is not available, the recipient may be the source of the NK cells.
* HLA typing will be performed by the Arkansas Children's Hospital clinical laboratory.
* If the recipient expresses HLA-C group I, HLA-C group II, and Bw4 KIR ligands, then a KIR-ligand mismatched haploidentical donor cannot be found, and the recipient will be the source of the NK cells.
* If the recipient fails to express one or more of the primary KIR ligands (HLA-C group I, HLA-C group II, and Bw4) then family member donors will be HLA typed in an effort to find a haploidentical donor. If multiple haploidentical donors are available, KIR phenotyping will be performed in Dr. van Rhee's research laboratory to select a KIR mismatched donor whenever possible.
* Donor selection will be performed by the PI or one of the MD co-investigators if Dr. van Rhee is not available.
* Signed IRB approved consent and HIPAA authorization form.
* Donor is not HIV I/II (+).
* Donor is not HTLV-I/II (+).
* Donor is not Hepatitis B or C (+) unless positive due to previous vaccination or has received therapy and is negative for Hepatitis B or C by RT-PCR.
* Donor is a suitable candidate for insertion of apheresis catheter. Donors with unusual anatomy or vascular anomalies preventing insertion of a pheresis catheter will be rejected.
* Age 18 years or greater or has signed an Assent and be age ≥16 years.
* Donor has a negative pregnancy test by serum or urine test.
* In preparation for the peripheral blood mononuclear cell donation, the donor will undergo a detailed medical history and physical examination. Clinical studies will include blood chemistries (electrolytes, liver function and CRP) CBC with differential and platelets, PT/PTT, viral panel, EKG (age over 40 yrs), and chest x-ray (age over 40yrs). Fitness to donate cells for NK expansion will be evaluated by a physician not involved in the initial assessment of the exp-NK cell recipient for enrollment onto the protocol.
* Serologic evaluation will be used to assess exposure to syphilis, West Nile Virus, Chagas, CMV IgG, hepatitis B, and C, HIV I and II, and HTLV I/II. An HIV-I/II[+] and HTLV-1/II (+) donor will be rejected on medical grounds. Donors who been vaccinated against hepatitis B and who have antibodies against hepatitis B surface antigen are allowed.
* Haplo-identical donor must not have prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has not received treatment for one year prior to donation.

Exclusion Criteria:

* Patient (Recipient of NK Cells) Exclusion criteria
* History of poorly controlled hypertension, diabetes mellitus, or any other serious medical illness or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol or could be considered to be an exclusion criterion deemed by the PI.
* Patients must not have prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has not received treatment for one year prior to enrollment. Other cancers will only be acceptable if the patient's life expectancy exceeds three years as determined by the PI.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of registration. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frits van Rhee, M.D., PHD., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Treatment: Bortezomib (1.0 mg/m2, IV) Days -9,-6,-2 (3 doses) Mesna (30 mg/kg, IV) Days -7, -6 (2 doses) Cyclophasphamide (60 mg/kg, IV) Day -7 (1 dose) Dexamethasone (40 mg, PO) Days -6 to -3 (4 doses) Expanded Natural Killer (exp-NK) Cell Infusion Day 0 (1 dose) Aldesleukin (IL-2) (3x10^6 IU, SC) Days 0 to 12 (13 doses)
Period: Overall Study
Arm/Group | Study Treatment
Started | 10
Completed | 8
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Study Treatment
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Efficacy
Description: Number of participants with an objective response of Partial Response (PR) or better according to European Society for Blood and Marrow Transplantation (EBMT) criteria within 180 days post Expanded Natural Killer Cell Infusion. The minimum criteria to meet the EBMT definition of PR or better included: >= 50% reduction in size of soft tissue plasmacytomas (if assessed); AND >= 50% reduction in plasma cells in bone marrow biopsy (if biopsy was performed and if >= 30% plasma cells at baseline); AND >=50% reduction in serum M protein and reduction in urine M protein >= 90% or to 200 mg/24hr OR >= 50% decrease in the difference between involved and uninvolved serum free light chain levels (if serum M protein < 1 g/dL, urine < 200 mg/24 hrs, and an involved serum free light chain level >= 10 mg/dL at baseline).
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Groups:
- Velcade for Anti-MM Therapy: Day(s) -9,-6,-2 3 doses of Bortezomib at 1.0 mg/m2, i.v.
  Bortezomib: bortezomib given days -9, -6, and -2 at 1.0mg/m2, i.v.
Arm/Group | Velcade for Anti-MM Therapy
Number analyzed (Participants) | 8
Participants | 1

ADVERSE EVENTS:
Time Frame: Data were collected from initiation of study therapy through 180 days post expanded natural killer cell infusion.
Arm/Group | Study Treatment
All-Cause Mortality (participants affected / at risk) | 3/8
Serious Adverse Events (participants affected / at risk) | 6/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Treatment (N=8)
Grade 4 Anemia (Blood and lymphatic system disorders) | 1
Grade 4 Thrombocytopenia (Blood and lymphatic system disorders) | 6
Grade 4 Leukopenia (Blood and lymphatic system disorders) | 6
Grade 3 Constitutional Symptoms - Other (General disorders) | 1
Grade 2 Fever (General disorders) | 1
Grade 2 Rigors/Chills (General disorders) | 1
Grade 3 Skin Rash (Skin and subcutaneous tissue disorders) | 1
Grade 3 Diarrhea (Gastrointestinal disorders) | 1
Grade 3 Mucositis/Stomatitis (Gastrointestinal disorders) | 1
Grade 2 Nausea (Gastrointestinal disorders) | 1
Grade 5 Sepsis (Infections and infestations) | 1
Grade 3 Infection - other (Infections and infestations) | 1
Grade 5 Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Treatment (N=8)
Grade 1 Rhinitis (Immune system disorders) | 1
Grade 2 Rhinitis (Immune system disorders) | 1
Grade 1 Anemia (Blood and lymphatic system disorders) | 7
Grade 2 Anemia (Blood and lymphatic system disorders) | 8
Grade 3 Anemia (Blood and lymphatic system disorders) | 6
Grade 1 Blood - Other (Blood and lymphatic system disorders) | 1
Grade 2 Blood - Other (Blood and lymphatic system disorders) | 1
Grade 1 Thrombocytopenia (Blood and lymphatic system disorders) | 4
Grade 2 Thrombocytopenia (Blood and lymphatic system disorders) | 5
Grade 3 Thrombocytopenia (Blood and lymphatic system disorders) | 7
Grade 2 Leukopenia (Blood and lymphatic system disorders) | 8
Grade 3 Leukopenia (Blood and lymphatic system disorders) | 7
Grade 2 Cardiac General - Other (Cardiac disorders) | 1
Grade 2 Hypotension (Cardiac disorders) | 1
Grade 1 Fatigue (General disorders) | 3
Grade 2 Fatigue (General disorders) | 4
Grade 1 Fever (General disorders) | 3
Grade 2 Fever (General disorders) | 2
Grade 1 Rigors/Chills (General disorders) | 3
Grade 2 Rigors/Chills (General disorders) | 1
Grade 1 Sweating (General disorders) | 1
Grade 1 Weight Loss (General disorders) | 1
Grade 1 Alopecia (Skin and subcutaneous tissue disorders) | 1
Grade 2 Alopecia (Skin and subcutaneous tissue disorders) | 1
Grade 1 Dermatology - Other (Skin and subcutaneous tissue disorders) | 1
Grade 2 Dermatology - Other (Skin and subcutaneous tissue disorders) | 1
Grade 2 Dry Skin (Skin and subcutaneous tissue disorders) | 1
Grade 1 Skin Rash (Skin and subcutaneous tissue disorders) | 1
Grade 2 Hypothyroidism (Endocrine disorders) | 1
Grade 1 Anorexia (Gastrointestinal disorders) | 1
Grade 2 Anorexia (Gastrointestinal disorders) | 1
Grade 1 Diarrhea (Gastrointestinal disorders) | 3
Grade 2 Diarrhea (Gastrointestinal disorders) | 2
Grade 1 Dry Mouth (Gastrointestinal disorders) | 1
Grade 1 Nausea (Gastrointestinal disorders) | 5
Grade 2 Nausea (Gastrointestinal disorders) | 1
Grade 1 Alkaline Phosphatase Increase (Hepatobiliary disorders) | 4
Grade 1 Bilirubin Increase (Hepatobiliary disorders) | 3
Grade 2 Bilirubin Increase (Hepatobiliary disorders) | 2
Grade 3 Bilirubin Increase (Hepatobiliary disorders) | 1
Grade 1 Hypoalbuminemia (Hepatobiliary disorders) | 7
Grade 2 Hypoalbuminemia (Hepatobiliary disorders) | 6
Grade 1 SGOT (AST) Increase (Hepatobiliary disorders) | 4
Grade 2 SGOT (AST) Increase (Hepatobiliary disorders) | 1
Grade 4 SGOT (AST) Increase (Hepatobiliary disorders) | 1
Grade 1 SGPT (ALT) Increase (Hepatobiliary disorders) | 3
Grade 2 SGPT (ALT) Increase (Hepatobiliary disorders) | 1
Grade 3 SGPT (ALT) Increase (Hepatobiliary disorders) | 1
Grade 4 SGPT (ALT) Increase (Hepatobiliary disorders) | 1
Grade 3 Febrile Neutropenia (Infections and infestations) | 1
Grade 3 Urinary Tract Infection (Infections and infestations) | 1
Grade 2 Pneumonia (Infections and infestations) | 1
Grade 2 Edema - Trunk/Genital (Blood and lymphatic system disorders) | 1
Grade 1 Bicarbonate Decrease (Metabolism and nutrition disorders) | 5
Grade 2 Bicarbonate Decrease (Metabolism and nutrition disorders) | 2
Grade 3 Bicarbonate Disease (Metabolism and nutrition disorders) | 1
Grade 1 Hyperglycemia (Metabolism and nutrition disorders) | 7
Grade 2 Hyperglycemia (Metabolism and nutrition disorders) | 5
Grade 3 Hyperglycemia (Metabolism and nutrition disorders) | 1
Grade 1 Hyperkalemia (Metabolism and nutrition disorders) | 2
Grade 2 Hyperkalemia (Metabolism and nutrition disorders) | 1
Grade 3 Hyperkalemia (Metabolism and nutrition disorders) | 1
Grade 1 Hypermagnesemia (Metabolism and nutrition disorders) | 6
Grade 3 Hypermagnesemia (Metabolism and nutrition disorders) | 1
Grade 1 Hypernatremia (Metabolism and nutrition disorders) | 1
Grade 2 Hypocalcemia (Metabolism and nutrition disorders) | 7
Grade 3 Hypocalcemia (Metabolism and nutrition disorders) | 3
Grade 4 Hypocalcemia (Metabolism and nutrition disorders) | 2
Grade 1 Hypokalemia (Metabolism and nutrition disorders) | 7
Grade 3 Hypokalemia (Metabolism and nutrition disorders) | 1
Grade 1 Hypomagnesemia (Metabolism and nutrition disorders) | 2
Grade 2 Hypomagnesemia (Metabolism and nutrition disorders) | 1
Grade 1 Hyponatremia (Metabolism and nutrition disorders) | 7
Grade 3 Hyponatremia (Metabolism and nutrition disorders) | 3
Grade 1 Hypophosphatemia (Metabolism and nutrition disorders) | 4
Grade 2 Hypophosphatemia (Metabolism and nutrition disorders) | 7
Grade 3 Hypophosphatemia (Metabolism and nutrition disorders) | 6
Grade 4 Hypophosphatemia (Metabolism and nutrition disorders) | 1
Grade 1 Gait/Walking (Musculoskeletal and connective tissue disorders) | 1
Grade 2 Muscle Weakness: Whole Body (Musculoskeletal and connective tissue disorders) | 4
Grade 3 Muscle Weakness: Whole Body (Musculoskeletal and connective tissue disorders) | 1
Grade 1 Confusion (Psychiatric disorders) | 2
Grade 2 Confusion (Psychiatric disorders) | 1
Grade 3 Confusion (Psychiatric disorders) | 1
Grade 4 Confusion (Psychiatric disorders) | 1
Grade 1 Dizziness (General disorders) | 2
Grade 1 Memory Impairment (Psychiatric disorders) | 1
Grade 1 Mood Alteration (Psychiatric disorders) | 2
Grade 2 Mood Alteration (Psychiatric disorders) | 2
Grade 1 Sensory Neuropathy (Nervous system disorders) | 2
Grade 2 Sensory Neuropathy (Nervous system disorders) | 2
Grade 3 Pain: Abdomen - NOS (General disorders) | 1
Grade 1 Headache (General disorders) | 1
Grade 2 Pain: Joint (Musculoskeletal and connective tissue disorders) | 1
Grade 1 Pain: Lower Back (Musculoskeletal and connective tissue disorders) | 2
Grade 2 Pain: Middle Back (Musculoskeletal and connective tissue disorders) | 1
Grade 1 Pain - NOS (General disorders) | 1
Grade 2 Pain: Upper Back (Musculoskeletal and connective tissue disorders) | 1
Grade 2 Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Grade 1 Cough (Respiratory, thoracic and mediastinal disorders) | 4
Grade 2 Cough (Respiratory, thoracic and mediastinal disorders) | 1
Grade 1 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Grade 2 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Grade 3 Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Grade 1 Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 1
Grade 2 Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 1
Grade 1 Creatinine Increase (Renal and urinary disorders) | 4
Grade 2 Creatinine Increase (Renal and urinary disorders) | 2
Grade 2 Thrombosis/Embolism (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes